CLINICAL TRIAL: NCT00365261
Title: Effect of Eszopiclone (Lunesta) on Sleep Disturbance and Pain in Cancer
Brief Title: Effect of Eszopiclone on Sleep Disturbance and Pain in Cancer
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University of California, San Diego (Other)
Responsible Party: Principal Investigator, Joel E. Dimsdale, M.D., Professor, University of California, San Diego
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: UCSD 060340; ESRC 054 (Other: Sepracor)
Record Dates: First submitted 2006-08-15; First posted 2006-08-17 (Estimated); Results first posted 2011-09-29 (Estimated); Last update posted 2016-07-11 (Estimated); Status verified 2016-06

CONDITIONS: Sleep Initiation and Maintenance Disorders
Keywords: pain; fatigue; sleep; bone marrow transplant; cancer
MeSH Terms: conditions — Sleep Initiation and Maintenance Disorders; Pain; Fatigue; Neoplasms | interventions — Eszopiclone

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- eszopiclone (Active Comparator): active drug
  Interventions: Drug: Eszopiclone
- placebo (Placebo Comparator): placebo
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Eszopiclone — eszopiclone 2 to 3 mg po at bedtime
  Other Names: Lunesta
  Arms: eszopiclone
Drug: Placebo — placebo 2 to 3 mg po at bedtime
  Arms: placebo

SUMMARY:
To assess the effectiveness of Lunesta on cancer patients who have received chemotherapy and who require patient controlled analgesia (PCA), specifically to assess whether Lunesta will:

* improve sleep thereby decreasing need for opiates via PCA
* improve sleep thereby decreasing pain by self report
* improve sleep thereby decreasing fatigue by self report

DETAILED DESCRIPTION:
Pain and fatigue are the most common symptom complaints of cancer patients. Although dramatic improvements have come about in recognizing and treating cancer related pain, less progress has been made in treating fatigue. Interventions to improve sleep may offer benefit in terms of pain and fatigue.

One of the less commonly recognized side effects of opiate use is sleep disruption.

Experimentally-induced sleep disruption lowers the threshold for detection of painful stimuli. Thus, although opiates are obviously helpful for pain, they do so at certain "costs": they increase next day fatigue, constipation, and have other side effects; they disrupt sleep which further increases next day fatigue; and finally, by virtue of their sleep disruptive properties, they lower the threshold for pain stimuli.

Cancer patients requiring chemotherapy commonly require PCA because of oral mucositis. The objective of this study is to assess whether opiate usage may be reduced and complaints of fatigue and pain be lessened if patients had better sleep.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female patients hospitalized for chemotherapy or blood/bone marrow transplant.
2. Age 20 - 75
3. Not currently regularly taking any prescribed sleeping pill more often than 4x/week.
4. Can tolerate oral medication.

Exclusion Criteria:

1. Patients with a current history of substance abuse
2. Patients with a history of allergic response to Lunesta.
3. Patient who require additional oral or parenteral opioids after starting PCA opioid treatment.

Ages: 20 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 45 (Actual)
Dates: Start 2006-09; Primary Completion 2009-12 (Actual); Study Completion 2009-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Joel E Dimsdale, MD, Principal Investigator — UCSD
Locations (1):
- UCSD Thornton Hospital, La Jolla, California, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Dimsdale JE, Ball ED, Carrier E, Wallace M, Holman P, Mulroney C, Shaikh F, Natarajan L. Effect of eszopiclone on sleep, fatigue, and pain in patients with mucositis associated with hematologic malignancies. Support Care Cancer. 2011 Dec;19(12):2015-20. doi: 10.1007/s00520-010-1052-1. Epub 2010 Nov 30. PMID 21116652

RESULTS

PARTICIPANT FLOW:
Groups:
- Eszopiclone: receipt of active drug
- Placebo: receipt of placebo
Period: Overall Study
Arm/Group | Eszopiclone | Placebo
Started | 23 | 22
Completed | 20 | 19
Not Completed | 3 | 3

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Eszopiclone | Placebo | Total
Number analyzed (Participants) | 23 | 22 | 45
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 23 | 20 | 43
  >=65 years | 0 | 2 | 2
Age, Continuous [Mean (Standard Deviation); unit: years] | 45.52 (13.06) | 46 (15.86) | 45.76 (14.33)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 13 | 9 | 22
  Male | 10 | 13 | 23
Region of Enrollment [Number; unit: participants]
  United States | 23 | 22 | 45

OUTCOME MEASURES:

1. Primary Outcome: Pain
Description: Pain was assessed with a 10-cm visual analog scale (0 = "no pain at all"; 10 = "severe, uncontrolled pain").
Time Frame: post dosing
Measure: Mean (Standard Error); unit: scores on a scale
Arm/Group | Eszopiclone | Placebo
Number analyzed (Participants) | 23 | 22
scores on a scale | 3.72 (0.38) | 5.41 (0.47)

2. Primary Outcome: Patient Self-report Data on Fatigue
Description: Patients completed the five-item Profile of Mood States Scale, Short Form (POMS-SF) Fatigue-Inertia Scale to rate their fatigue complaints (scores range from 0 to 28; higher scores denote more fatigue).
Time Frame: 2 days post treatment
Measure: Mean (Standard Error); unit: scores on a scale
Arm/Group | Eszopiclone | Placebo
Number analyzed (Participants) | 23 | 22
scores on a scale | 2.41 (0.20) | 2.77 (0.17)

3. Secondary Outcome: Opiate Dosing From Patient Controlled Analgesia
Description: Morphine or dilaudid dose delivered at fixed rate with optional self-administered prn boluses. Dilaudid doses were converted into morphine equivalents by multiplying the dose by 5.
Time Frame: 2 days post dosing
Measure: Median (Inter-Quartile Range); unit: mg
Arm/Group | Eszopiclone | Placebo
Number analyzed (Participants) | 23 | 22
mg | 36.35 [17.57 to 58.46] | 40.94 [23.37 to 66.19]

ADVERSE EVENTS:
Arm/Group | Eszopiclone | Placebo
Serious Adverse Events (participants affected / at risk) | 0/23 | 0/22
Other Adverse Events (participants affected / at risk) | 3/23 | 3/22
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Eszopiclone (N=23) | Placebo (N=22)
fatigue (General disorders) | 3 (3) | 3 (3) — fatigue or drowsiness

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No